CLINICAL TRIAL: NCT05514483
Title: Effect of a 5-HT3 Receptor Antagonist on Respiratory Drive in Spontaneously Breathing Mechanically Ventilated Patients With Acute Respiratory Distress Syndrome (ARDS): a Pilot Proof-of-concept Crossover Non-randomized Controlled Trial
Brief Title: 5-HT3 Receptor Antagonist and Respiratory Drive in Patients With ARDS
Acronym: DRIVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Yiorgos Alexandros Cavayas, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-2502
Record Dates: First submitted 2022-08-17; First posted 2022-08-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Ondansetron
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Sodium Chloride; Saline Solution; Ondansetron

STUDY DESIGN:
Intervention Model Description: Non-randomized crossover controlled trial with two interventions and one sequence. The sequence of treatment is first placebo and secondly ondansetron.
Masking Description: Because of the single sequence of administration, blinding of study personnel would not be possible. As the primary outcome is a continuously electronically recorded physiological parameter that does not require any human interpretation, single blinding should not result in any observation bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): All participants will receive a single injection of placebo, followed, three hours later, by a single injection of ondansetron.
  Interventions: Drug: Placebo
- Ondansetron (Active Comparator): All participants will receive a single injection of placebo, followed, three hours later, by a single injection of ondansetron.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Placebo — Single intravenous dose of 10 mL of sodium chloride (NaCl) 0.9% over 15 minutes.
  Other Names: NaCl 0.9%; Normal Saline; Sodium chloride
  Arms: Placebo
Drug: Ondansetron — Single intravenous dose of ondansetron hydrochloride dihydrate 0.15 mg/kg (maximum 16 mg) in 10 mL of NaCl 0.9% over 15 minutes.
  Other Names: Ondansetron hydrochloride dihydrate
  Arms: Ondansetron

SUMMARY:
This is a pilot study aimed at acquiring primary physiological data, describing and estimating the effects of a 5-HT3 receptor antagonist (ondansetron) on respiratory drive in patients with acute respiratory distress syndrome (ARDS). The results of this study will determine the interest and feasibility of assessing the clinical applications of ondansetron in reducing patient self-inflicted lung injury (P-SILI) in ARDS, in subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18-75 years old)
* Berlin Criteria for Acute Respiratory Distress Syndrome (ARDS) (1):

  * Hypoxemic respiratory failure with a patrial pressure of arterial oxygen to fraction of inspired oxygen ratio (PaO2:FiO2 ratio) < 300
  * Bilateral opacities not fully explained by effusions, lung/lobar collapse, or nodules on chest imaging that appeared within 7 days of a known clinical insult
  * Respiratory failure not fully explained by cardiac failure or fluid overload
* Has been mechanically ventilated > 48 hours
* Planned to remain mechanically ventilated for the next 24 hours
* Currently on Pressure Support Ventilation or planning to go on pressure support ventilation in the next 24 hours

Exclusion Criteria:

* Having received a 5-HT3 antagonist in the last 24 hours, or planning to use one in the next 24 hours
* Recently treated for bleeding varices, stricture, hematemesis, esophageal trauma, recent esophageal surgery or other contraindication for nasogastric tube placement
* Severe coagulopathy (platelet count< 10 000 or International Normalized Ratio (INR) > 3)
* Neuromuscular disease that impairs ability to ventilate spontaneously (including C5 or higher spinal cord injury, amyotrophic lateral sclerosis, Guillain-Barre syndrome or myasthenia gravis)
* Treating clinician refusal, or unwillingness to commit to pressure support ventilation for at least 6 hours.
* Pregnancy
* Liver cirrhosis (Child B or C) or other severe impairment of hepatic function
* Congestive heart failure
* Bradyarrhythmia (baseline pulse<55/min)
* Known long QT syndrome
* QTc prolongation>450 msec, noted on prior or screening ECG, or who are taking medication known to cause QT prolongation
* Hypersensitivity or other known intolerance to ondansetron or other 5-HT3 antagonists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-03-06 (Estimated); Study Completion 2024-05-06 (Estimated)

PRIMARY OUTCOMES:
Pressure-time product of the esophageal pressure per minute | Continuous measurement during each 2-hour phase
  Difference in mean pressure-time product of the esophageal pressure per minute between placebo phase and ondansetron phase

SECONDARY OUTCOMES:
Respiratory rate | Continuous measurement during each 2-hour phase
  Difference in mean respiratory rate between placebo phase and ondansetron phase
Tidal volume | Continuous measurement during each 2-hour phase
  Difference in mean tidal volume between placebo phase and ondansetron phase
Pressure-time product of the esophageal pressure per breath | Continuous measurement during each 2-hour phase
  Difference in mean pressure-time product of the esophageal pressure per breath between placebo phase and ondansetron phase
Esophageal pressure swings | Continuous measurement during each 2-hour phase
  Difference in mean esophageal pressure swings between placebo phase and ondansetron phase
Transpulmonary pressure swings | Continuous measurement during each 2-hour phase
  Difference in mean transpulmonary pressure swings between placebo phase and ondansetron phase
Estimated occlusion pressure at 0.1 msec (P0.1) | Continuous measurement during each 2-hour phase
  Difference in mean estimated occlusion pressure at 0.1 msec (P0.1) between placebo phase and ondansetron phase
Peak electrical activity of the diaphragm (Eadi) | Continuous measurement during each 2-hour phase
  Difference in mean peak Eadi between placebo phase and ondansetron phase
Area under the Eadi curve | Continuous measurement during each 2-hour phase
  Difference in area under the Eadi curve between placebo phase and ondansetron phase
End-tidal CO2 (EtCO2) | Continuous measurement during each 2-hour phase
  Difference in mean EtCO2 between placebo phase and ondansetron phase
Volume of expired CO2 (VCO2) | Continuous measurement during each 2-hour phase
  Difference in mean VCO2 between placebo phase and ondansetron phase
Oxygen saturation estimated by pulse oximetry (SpO2) | Measurement every 5 minutes during each 2-hour phase
  Difference in mean SpO2 between placebo phase and ondansetron phase
Partial pressure of carbon dioxide in arterial blood (PaCO2) | Measurement every 30 minutes during each 2-hour phase
  Difference in mean PaCO2 between placebo phase and ondansetron phase
Partial pressure of oxygen in arterial blood (PaO2) | Measurement every 30 minutes during each 2-hour phase
  Difference in mean PaO2 between placebo phase and ondansetron phase
Heart rate | Measurement every 5 minutes during each 2-hour phase
  Difference in mean heart rate between placebo phase and ondansetron phase
Mean arterial pressure (MAP) | Measurement every 5 minutes during each 2-hour phase
  Difference in mean MAP between placebo phase and ondansetron phase
Corrected QT length (QTc) | Measurement once (at the 1 hour-mark) during each 2-hour phase
  Difference in QTc between placebo phase and ondansetron phase
Temperature | Hourly measurement during each 2-hour phase
  Difference in mean temperature between placebo phase and ondansetron phase
Richmond Agitation and Sedation Scale (RASS) | Hourly measurement during each 2-hour phase
  Difference in mean Richmond Agitation and Sedation Scale (RASS) between placebo phase and ondansetron phase. This scale goes from -5 (unraousable) to +4 (combative).
Critical care Pain Observation Tool (CPOT) | Hourly measurement during each 2-hour phase
  Difference in mean Critical care Pain Observation Tool (CPOT) between placebo phase and ondansetron phase. This scale goes from 0 (lowest pain level) to 10 (highest pain level).

OTHER OUTCOMES:
Enrolment | Monthly through study completion (estimated 6 months)
  Number of eligible patients and enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yiorgos Alexandros Cavayas, MD MSc FRCPC, Principal Investigator — Hopital du Sacré Coeur de Montréal, Centre de recherche du centre intégré universitaire de santé et services sociaux du Nord-de-l'Ile-de-Montréal
Locations (1):
- Hôpital Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No